CLINICAL TRIAL: NCT06972446
Title: A Phase 2, Multicenter, Platform Study of Targeted Therapies for the Treatment of Adult Subjects With Moderately to Severely Active Rheumatoid Arthritis
Brief Title: A Study to Evaluate Different Targeted Therapies for Patients With Rheumatoid Arthritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M25-056; 2025-520721-21-00 (Other: EU CT)
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — lutikizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Substudy 1: Lutikizumab Monotherapy (Experimental): Participants will be randomized to initially receive Lutikizumab Dose A followed by Lutikizumab Dose B
  Interventions: Drug: Lutikizumab
- Substudy 1: Matching Placebo Monotherapy (Placebo Comparator): Participants will be randomized to receive a matching placebo dose equivalent to the Lutikizumab monotherapy.
  Interventions: Drug: Placebo
- Substudy 2: Ravagalimab Monotherapy (Experimental): Participants will be randomized to receive Ravagalimab
  Interventions: Drug: Ravagalimab
- Substudy 2: Matching Placebo Monotherapy (Placebo Comparator): Participants will be randomized to receive a matching placebo dose equivalent to the Ravagalimab monotherapy
  Interventions: Drug: Placebo
- SubStudy 3: Lutikizumab and Ravagalimab Combination Therapy (Experimental): Participants will be randomized to be administered Lutikizumab and Ravagalimab doses
  Interventions: Drug: Lutikizumab; Drug: Ravagalimab
- Substudy 3: Matching Placebo Combination Therapy (Placebo Comparator): Participants will be randomized to receive matching placebo doses equivalent to the Lutikizumab and Ravagalimab combination therapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lutikizumab — Subcutaneous (SC) injection
  Arms: SubStudy 3: Lutikizumab and Ravagalimab Combination Therapy; Substudy 1: Lutikizumab Monotherapy
Drug: Placebo — Subcutaneous (SC) injection
  Arms: Substudy 1: Matching Placebo Monotherapy; Substudy 2: Matching Placebo Monotherapy; Substudy 3: Matching Placebo Combination Therapy
Drug: Ravagalimab — Subcutaneous (SC) injection
  Arms: SubStudy 3: Lutikizumab and Ravagalimab Combination Therapy; Substudy 2: Ravagalimab Monotherapy

SUMMARY:
Rheumatoid Arthritis (RA) is a chronic inflammatory disease causing pain, stiffness, swelling and loss of joint function. This study will evaluate the efficacy and safety of targeted therapies through a series of substudies for the treatment of moderately to severely active Rheumatoid Arthritis (RA).

This study currently includes 3 substudies evaluating different treatments in participants with RA. Substudy 1 will evaluate lutikizumab monotherapy (treatment given alone) compared to placebo (looks like the study treatment but contains no medicine). Substudy 2 will evaluate ravagalimab monotherapy compared to placebo and Substudy 3 will evaluate lutikizumab and ravagalimab combination therapy (treatments given together) compared to placebo. Approximately 180 participants who have failed 1 or 2 biologic/targeted synthetic disease-modifying antirheumatic drug (tsDMARD) therapies will be enrolled in the study at approximately 65 sites worldwide.

There may be higher treatment burden for participants in this trial compared to their standard of care treatment without participating in this study. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* At any time prior to the Screening Visit, participant must have been treated for > or = 3 months with at least 1 b/tsDMARD therapy but continued to exhibit active RA, or had to discontinue due to intolerability or toxicity, irrespective of treatment duration. The maximum cap for prior use of b/tsDMARD is 2.
* Participant must be on a stable dose of methotrexate (MTX)

Exclusion Criteria:

* Participant is taking nonsteroidal anti-inflammatory drugs (NSAIDs), acetaminophen/paracetamol, low-potency opioids (tramadol, codeine, hydrocodone, alone or in combination with acetaminophen), oral corticosteroids (equivalent to ≤ 10 mg/day of prednisone), or inhaled corticosteroids for stable medical conditions unless they have been on stable doses for ≥ 1 week prior to Baseline Visit.
* History of any arthritis with onset prior to age 17 years or current diagnosis of inflammatory joint disease other than rheumatoid arthritis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With an American College of Rheumatology 50% (ACR50) Response | At Week 12
  Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR50 response criteria:
  1. ≥ 50% improvement in 68-tender joint count;
  2. ≥ 50% improvement in 66-swollen joint count; and
  3. ≥ 50% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP)
Number of Participants with Adverse Events (AEs) | Up to Approximately Week 22
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response | At Week 12
  Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR20 response criteria:
  1. ≥ 20% improvement in 68-tender joint count;
  2. ≥ 20% improvement in 66-swollen joint count; and
  3. ≥ 20% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP)
Percentage of Participants With an American College of Rheumatology 70% (ACR70) Response | At Week 12
  Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR70 response criteria:
  1. ≥ 70% improvement in 68-tender joint count;
  2. ≥ 70% improvement in 66-swollen joint count; and
  3. ≥ 70% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP)
Percentage Of Participants Achieving Low Disease Activity (LDA) per Disease Activity Score-28 With C-Reactive Protein (DAS28-CRP) | At Week 12
  The Disease Activity Score (DAS) 28 is a validated index of rheumatoid arthritis disease activity. Scores on the DAS28 range from 0 (lowest disease activity) to 10 (highest disease activity). LDA is defined as a score of < or = to 3.2.
Percentage Of Participants Achieving Clinical Remission (CR) per DAS28 (CRP) | At Week 12
  The Disease Activity Score (DAS) 28 is a validated index of rheumatoid arthritis disease activity. Scores on the DAS28 range from 0 (lowest disease activity) to 10 (highest disease activity). CR remission is defined as a score of less than 2.6
Change from Baseline in DAS28 (CRP) | At Week 12
  The DAS28-CRP is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (NRS), and high-sensitivity C-reactive protein (hsCRP; in mg/L). Scores on the DAS28-CRP range from 0 to approximately 10, where higher scores indicate more disease activity.
Percentage Of Participants Achieving LDA per Clinical Disease Activity Index (CDAI) | At Week 12
  The CDAI is a composite index for assessing disease activity. The total CDAI score ranges from 0 to 21 with higher scores indicating higher disease activity. LDA is defined as a score from 2.8 to ≤ 10.
Percentage Of Participants Achieving CR per CDAI | At Week 12
  The CDAI is a composite index for assessing disease activity. The total CDAI score ranges from 0 to 21 with higher scores indicating higher disease activity. CR remission is defined as a score of less than 2.8

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (54):
- United States (35):
  - Sun Valley Arthritis Center /ID# 278331, Peoria, Arizona
  - Private Practice - Dr. David S. Hallegua /ID# 277608, Beverly Hills, California
  - Advanced Clinical Research Center, LLC dba TriWest Research Associates /ID# 277826, Chula Vista, California
  - Newport Huntington Medical Group /ID# 272439, Huntington Beach, California
  - Cohen Medical Centers /ID# 278341, Thousand Oaks, California
  - Inland Rheumatology & Osteoporosis Medical Group /ID# 272449, Upland, California
  - Tekton Research - Fort Collins - East Harmony Road /ID# 272472, Fort Collins, Colorado
  - Highlands Advanced Rheumatology And Arthritis Center - Avon Park /ID# 272298, Avon Park, Florida
  - Clinical Research Of West Florida - Phase I Unit /ID# 272428, Clearwater, Florida
  - Neoclinical Research - Hialeah /ID# 272070, Hialeah, Florida
  - Swati Shah, MD Rheumatology /ID# 273624, Jacksonville, Florida
  - Life Clinical Trials /ID# 272589, Margate, Florida
  - HMD Research LLC /ID# 272432, Orlando, Florida
  - Clinical Research Of West Florida - Tampa - North Howard Avenue /ID# 272755, Tampa, Florida
  - Deerbrook Medical Associates /ID# 273439, Libertyville, Illinois
  - Willow Rheumatology and Wellness, PLLC /ID# 272691, Willowbrook, Illinois
  - Accurate Clinical Research (SMO/Network/Consortium) /ID# 272650, Lake Charles, Louisiana
  - AA Medical Research Center - Grand Blanc /ID# 272496, Grand Blanc, Michigan
  - Albuquerque Center For Rheumatology /ID# 272301, Albuquerque, New Mexico
  - Joint And Muscle Research Institute /ID# 277290, Charlotte, North Carolina
  - DJL Clinical Research, PLLC /ID# 272387, Charlotte, North Carolina
  - Paramount Medical Research and Consulting /ID# 272474, Middleburg Heights, Ohio
  - Altoona Center For Clinical Research /ID# 272479, Duncansville, Pennsylvania
  - Low Country Rheumatology /ID# 277607, Summerville, South Carolina
  - West Tennessee Research Institute /ID# 272453, Jackson, Tennessee
  - Arthritis & Rheumatology Research Institute /ID# 272299, Allen, Texas
  - Tekton Research - West Gate /ID# 272270, Austin, Texas
  - Trinity Universal Research Associates - Carrollton /ID# 272577, Carrollton, Texas
  - Arthritis Care Of Texas /ID# 277961, Corpus Christi, Texas
  - Accurate Clinical Research - Houston /ID# 272271, Houston, Texas
  - Private Practice - Dr. Laila A. Hassan /ID# 272297, Houston, Texas
  - Southwest Rheumatology Research /ID# 272268, Mesquite, Texas
  - Texas Rheumatology Research Institute Llc /Id# 278010, Plano, Texas
  - Epic Medical Research /ID# 272656, Red Oak, Texas
  - Dynamed Clinical Research - Tomball /ID# 272452, Tomball, Texas
- Canada (2):
  - Care Clinic - Calgary /ID# 274405, Calgary, Alberta
  - Dr. Latha Naik Medical Professional Corporation /ID# 274403, Saskatoon, Saskatchewan
- MEDICAL PLUS Research s.r.o /ID# 271926, Uherské Hradiště, Czechia
- Germany (4):
  - Rheumateam Lahn-Dill-Siegerland /ID# 274858, Wetzlar, Hesse
  - Universitaetsklinikum Bonn /ID# 272808, Bonn, North Rhine-Westphalia
  - Krankenhaus Porz Am Rhein /ID# 272903, Cologne, North Rhine-Westphalia
  - MVZ Rheumatologie und Autoimmunmedizin in Hamburg /ID# 272795, Hamburg
- Vital-Medicina Kft. /ID# 272858, Veszprém, Fejér, Hungary
- Puerto Rico (4):
  - Clinical Research Investigator Group, LLC /ID# 274821, Bayamón
  - Centro Reumatologico De Caguas /ID# 277918, Caguas
  - Reuviva Research Center, LLC /ID# 277140, Guaynabo
  - Santurce Clinical Trials and Infusion Center /ID# 277927, San Juan
- South Korea (4):
  - SoonChunHyang University Hospital Cheonan /ID# 277624, Cheonan-si, Chungcheongnam-do
  - Ajou University Hospital /ID# 273647, Suwon, Gyeonggido
  - Hanyang University Seoul Hospital /ID# 273625, Seoul, Seoul Teugbyeolsi
  - SMG-SNU Boramae Medical Center /ID# 273627, Seoul, Seoul Teugbyeolsi
- Spain (3):
  - Complejo Hospitalario Universitario A Coruña /ID# 272609, A Coruña, A Coruna
  - Hospital de Basurto /ID# 272610, Bilbao, Vizcaya
  - Consorci Hospital General Universitario de Valencia /ID# 272615, Valencia

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-056